CLINICAL TRIAL: NCT04103489
Title: Eculizumab in HELLP Syndrome
Brief Title: The Use of Eculizumab in HELLP Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00193549; 1K12HD085845-01 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: HELLP Syndrome (HELLP), Third Trimester; Complement Abnormality; Morbidity;Newborn; Maternal Injury; Preeclampsia Severe
MeSH Terms: conditions — HELLP Syndrome | interventions — eculizumab

STUDY DESIGN:
Intervention Model Description: This will be an open label, phase 1 clinical trial. The investigators will investigate if eculizumab halts or prevents worsening or HELLP syndrome in women at 23-28 weeks gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HELLP Syndrome at less than 30 weeks gestation (Experimental): Women diagnosed with HELLP syndrome at 23-30 weeks gestation will receive eculizumab.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Participants will receive eculizumab at diagnosis of HELLP syndrome. Participants will receive a maximum of 4 doses.
  Other Names: Soliris

SUMMARY:
This research study is being performed to see if women diagnosed with early preterm Hemolysis, Elevated Liver Enzymes, Low Platelets (HELLP) syndrome (estimated gestational ages of 23-30 weeks) benefit from a medication called eculizumab (ECU). This drug blocks a part of the immune system called complement. By blocking this part of the immune system, eculizumab may stop or reverse the progression of the HELLP syndrome disease. The investigators will also look to see if this drug is effective and benefits both the mother and fetus.

DETAILED DESCRIPTION:
Preeclampsia is a devastating multisystem disorder of pregnancy that manifests as hypertension with or without proteinuria and/or end organ damage caused by endothelial dysfunction and occurs in 3-5% of all pregnancies. Notably, preeclampsia accounts for 30% of all preterm deliveries, which results in neonatal intensive care unit admissions, increased health care cost, severe neonatal morbidity, and neonatal mortality. HELLP (hemolysis, elevated liver enzymes, and low platelets) syndrome is the most severe variant of this disorder, and affects approximately 0.1-0.2% of all pregnancies. Despite its prevalence, the cellular biology of HELLP syndrome is unclear resulting in supportive treatment regimens like fetal monitoring, steroids for fetal lung maturity, magnesium for seizure prophylaxis, management of hypertension and ultimately delivery that results in iatrogenic preterm birth.

Complement is an enzymatic cascade of approximately 50 proteins which are activated by the classic pathway of complement, the lectin pathway of complement, and the alternative pathway of complement (APC). While the classic pathway depends on antigen-antibody complexes (i.e., lupus) for activation, the APC is antibody independent and has various triggers including infection, trauma, and pregnancy.

The investigators' research lab created a novel functional assay, the modified Ham (mHam) assay, to diagnose highly morbid diseases of the APC such atypical hemolytic uremic syndrome (aHUS). Because of the phenotypic similarities of aHUS and HELLP syndrome the investigators' lab undertook a study to test women diagnosed with complete (classic) HELLP and partial (atypical) HELLP syndrome established by Tennessee and American College of Obstetrics and Gynecology (ACOG) criteria to observe if there was dysregulation and overactivation of the APC. The investigators found that most women with HELLP syndrome have APC upregulation; furthermore, it could be inhibited in vitro with anti-C5 monoclonal antibody. In addition, the investigators recently showed approximately 50% of women with HELLP syndrome have germline mutations associated with regulatory proteins of the APC 12. These are the same mutations associated with aHUS; further, 4 of the 5 women with germline mutations are positive by the mHam assay correlating genotype to phenotype. With the investigators' current data that HELLP syndrome is similar to aHUS, the investigators propose an open label clinical trial of ECU administration to women with HELLP syndrome at 23-30 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with HELLP syndrome less than 30 weeks gestation.

Exclusion Criteria:

Women with

* Disseminated intravascular coagulopathy
* Non-reassuring fetal status necessitating delivery
* Non-viable fetuses
* Stroke
* Fetal demise intra-utero
* Eclamptic seizure
* Known atypical hemolytic uremic syndrome
* Familial or acquired thrombocytopenia purpura
* Paroxysmal nocturnal hemoglobinuria
* Allergy to eculizumab will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Change in aspartate aminotransferase (AST) level | Baseline, 72 hours
  AST measured in units/L.
Change in alanine aminotransferase (ALT) | Baseline, 72 hours
  ALT measured in IU/L.
Change in lactate dehydrogenase levels (LDH) | Baseline, 72 hours
  LDH measured in units/L.

SECONDARY OUTCOMES:
Latency of pregnancy | Up to 7 days
  Latency of pregnancy measured in days after eculizumab administration
Maternal number of units of blood products transfused | Up to 7 days
  Blood products (packed red blood cells, fresh frozen plasma, platelets, cryoprecipitate) measured in units.
Maternal postpartum length of stay | Up to 36 days
  Postpartum length of stay, measured from delivery to time of discharge in days.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Vaught, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided